CLINICAL TRIAL: NCT01050608
Title: Real Time Deployment of Multimodal Personal Dispenser Hand Hygiene System in a Multidisciplinary Intensive Care Unit.
Brief Title: Evaluation of Body-worn Multimodal Hand Hygiene System. Impact on Health-Care Associated Infections
Acronym: Sprixx-ICU
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Harbor Medical Inc. (Industry)
Responsible Party: Matthew D. Koff M.D. M.S., Dartmouth-Hitchcock Medical Center
Other Study IDs: 20655-ICU extension
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Nosocomial Infection
Keywords: Alcohol Rub; Hand Hygiene; Provider Feedback; Health Care Associated Infections
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sprixx Device Group: Treatment group utilizing multimodal hand hygiene device
  Interventions: Device: Body worn alcohol gel dispenser; Drug: 62% ethanol based hand cleanser; Behavioral: Educational component with regard to teaching CDC guidelines; Behavioral: Provider and group feedback
- Standard Hand Hygiene Group: Utilizing wall mounted dispensers and CDC based guidelines.

INTERVENTIONS:
Device: Body worn alcohol gel dispenser — Records hand hygiene events of provider and tabulates on the group level.
  Groups: Sprixx Device Group
Drug: 62% ethanol based hand cleanser — CDC based guidelines with regard to utilization in the health care environment "the nest"
  Groups: Sprixx Device Group
Behavioral: Educational component with regard to teaching CDC guidelines — 12 minute education prior to deploying device for all providers.
  Groups: Sprixx Device Group
Behavioral: Provider and group feedback — Provide feedback with regard to expected hand hygiene goals to providers and reported anonymous group results based on recorded information.
  Groups: Sprixx Device Group

SUMMARY:
Evaluate the efficacy of a multimodal hand hygiene system in the intensive care unit environment and evaluate any impact on health care associated infections.

DETAILED DESCRIPTION:
Deploy and utilize a novel body worn hand hygiene system that incorporates provider and group specific feedback allowing hand hygiene to occur directly within the patient environment. We hypothesize that by improving provider hand hygiene we will reduce health-care associated infection rates.

ELIGIBILITY:
Inclusion Criteria:

* All ICU patients

Exclusion Criteria:

* Patient is not in an ICU at our Institution

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Intensive Care Unit Patients Multidisciplinary Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 2954 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Reduction in healthcare associated infections (CRBSI and VAP) | 2 years

SECONDARY OUTCOMES:
Time to infections Hospital mortality Length of stay | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D. Koff, M.D. M.S., Principal Investigator — Dartmouth-Hitchcock Medical Center; Randy L Loftus, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-HItchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Anesthesiology 2008; 109 A54 ASA Abstracts